CLINICAL TRIAL: NCT00686803
Title: A Single-Center, Single-Dose, Placebo-Controlled, Randomized, Double-Blind, Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered PL-3994 in Subjects With Controlled Hypertension
Brief Title: Safety Study of Subcutaneously Administered PL-3994 in Subjects With Controlled Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PL3994-003
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Hypertension
Keywords: hypertension; controlled hypertension; hypertensives
MeSH Terms: conditions — Hypertension | interventions — PL-3994

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- PL3994 Dose A (Experimental): PL3994 Dose A
  Interventions: Drug: PL3994
- PL3994 Dose B (Experimental): PL3994 Dose B
  Interventions: Drug: PL3994
- PL3994 Dose C (Experimental): PL3994 Dose C
  Interventions: Drug: PL3994
- PL3994 Dose D (Experimental): PL3994 Dose D
  Interventions: Drug: PL3994
- PL3994 Dose E (Experimental): PL3994 Dose E
  Interventions: Drug: PL3994
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PL3994 — Study drug
  Arms: PL3994 Dose A; PL3994 Dose B; PL3994 Dose C; PL3994 Dose D; PL3994 Dose E
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and pharmacokinetics of subcutaneous (SC) PL-3994, relative to placebo in subjects with controlled hypertension. Including in this evaluation is the effect PL3994 has on blood pressure.

DETAILED DESCRIPTION:
Uncontrolled hypertension, including both hypertensive urgency and hypertensive emergency, is commonly seen in emergency rooms and other urgent care settings. Current standards of care include intravenously administered drugs, which can be difficult to titrate and require ongoing monitoring. This study examines the effect of PL-3994 on patients with controlled hypertension who are receiving antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have had a diagnosis of essential hypertension for at least 1 year, per subject verbal history
* Subject must be on a stable dose of at least one, but not more than 3 antihypertensive medications for at least 3 months, per subject verbal history.
* Subject must have a systolic blood pressure at screening between 100 and 150 mmHg, and diastolic blood pressure must not exceed 105 mmHg.

Exclusion Criteria:

* Subject weight greater than 100 kg or less than 50 kg.
* Any significant medical condition or abnormal safety laboratory results which, in the judgement of the Investigator would place the subject at significant risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fischkoff, MD, Study Director — Palatin Technologies, Inc; Robert Jordan, Study Director — Palatin Technologies, Inc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initiation Date: 28 April 2008 Completion Date: 21 July 2008 Cohort 1: 6 subjects: PL-3994 0.3 µg/kg; 1 subject Placebo Cohort 2: 6 subjects: PL-3994 0.1 µg/kg; 1 subject Placebo Cohort 3: 6 subjects: PL-3994 0.3 µg/kg; 1 subject Placebo; Study stopped after Cohort 3.
Pre-assignment Details: Some results (i.e.Pharmacodynamic results) may include analyses only for the Evaluable Subjects population.The Evaluable Subjects population consisted of subjects who received study drug and who had no major protocol deviations that would have excluded the subject from analysis, and for whom calculations of PK or PD parameters were possible.
Groups:
- PL-3994 0.1 µg/kg: PL-3994 0.1 µg/kg
- PL-3994 0.3 µg/kg: PL-3994 0.3 µg/kg
Period: Overall Study
Arm/Group | PL-3994 0.1 µg/kg | PL-3994 0.3 µg/kg | Placebo
Started | 6 | 12 | 3
Completed | 6 | 12 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PL-3994 0.1 µg/kg | PL-3994 0.3 µg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 12 | 3 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 3 | 21
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (5.24) | 51.7 (5.42) | 59.3 (5.13) | 53.3 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 10
  Male | 3 | 7 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Subcutaneous (SC) PL-3994 Relative to Placebo in Subjects With Controlled Hypertension.
Description: The pharmacokinetic profile parameters for PL-3994 were calculated using a non compartmental approach.
  •Maximum concentration (Cmax)
  The subject numbers below are the evaluable subjects only. The Evaluable Subjects population consisted of subjects who received study drug and who had no major protocol deviations that would have excluded the subject from analysis, and for whom calculations of PK parameters were possible.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PL-3994 0.1 µg/kg | PL-3994 0.3 µg/kg | Placebo
Number analyzed (Participants) | 6 | 12 | 3
ng/mL | 0 (0) | 0.366 (0.0656) | 0 (0)

2. Primary Outcome: Pharmacodynamics as Measured by cGMP Levels.
Description: Pharmacodynamic parameters were calculated from the baseline-adjusted plasma cGMP level-time data using WinNonlin® 5.0.1. Actual sample times were used in the calculations. Baseline was the pre-dose levels of plasma cGMP at Visit 2 (Day 1): Emax
  The patient numbers below represent the evaluable subjects only. The Evaluable Subjects population consisted of subjects who received study drug and who had no major protocol deviations that would have excluded the subject from analysis, and for whom calculations of PD parameters were possible.
Time Frame: 24 hours
Measure: Median (Full Range); unit: ng/mL
Arm/Group | PL-3994 0.1 µg/kg | PL-3994 0.3 µg/kg | Placebo
Number analyzed (Participants) | 3 | 8 | 1
ng/mL | 0.996 [0.38 to 1.03] | 1.435 [0.87 to 4.26] | 0.676 [0.676 to 0.676]

ADVERSE EVENTS:
Arm/Group | PL-3994 0.1 µg/kg | PL-3994 0.3 µg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 6/12 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 4.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PL-3994 0.1 µg/kg (N=6) | PL-3994 0.3 µg/kg (N=12) | Placebo (N=3)
Dizziness (Nervous system disorders) | 0 | 4 | 1
headache (Nervous system disorders) | 0 | 2 | 1
somnolence (Nervous system disorders) | 0 | 1 | 1
nausea (Gastrointestinal disorders) | 0 | 2 | 0
dizziness postural (Nervous system disorders) | 0 | 1 | 0
fatigue (General disorders) | 0 | 1 | 0
feeling hot (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
vessel puncture site pain (General disorders) | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 1 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
musculoskelatal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
platelet count decreased (Investigations) | 0 | 0 | 1
depersonalization (Psychiatric disorders) | 0 | 1 | 0
urinary tract inflammation (Renal and urinary disorders) | 1 | 0 | 0
ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI was an employed by Palatin, as he was/is an employee of the CRO hired by Palatin to conduct the study. All confidentiality agreed upon between Palatin and the CRO applies.